CLINICAL TRIAL: NCT05255471
Title: Olaparib Beyond Progression Compared to Platinum Chemotherapy After Secondary Cytoreductive Surgery in Recurrent Ovarian Cancer Patients. The Phase III Randomized, Open Label MITO 35b Study: a Project of the MITO-MANGO Groups.
Brief Title: MITO 35B: Olaparib Beyond Progression Compared to Platinum Chemotherapy After Secondary Cytoreductive Surgery in Recurrent Ovarian Cancer Patients.
Acronym: MITO 35B
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITO35B/EudraCT:2021-000245-41
Record Dates: First submitted 2022-02-01; First posted 2022-02-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer
Keywords: Recurrent ovarian cancer; Olaparib; Chemotherapy; Secondary Cytoreductive Surgery
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olaparib (Experimental)
  Interventions: Drug: Olaparib
- Chemotherapy (Active Comparator)
  Interventions: Drug: Chemotherapy drug

INTERVENTIONS:
Drug: Olaparib — Olaparib 300 mg, film-coated tablets, twice daily PO, d1- 28 continuously
  Arms: Olaparib
Drug: Chemotherapy drug — Platinum-based chemotherapy at the Investigator's choice among the following regimens:
  * Carboplatin (AUC5) plus Pegylated Liposomal Doxorubicin (PLD) 30mg/m2 on day 1 every 28 days for a maximum of 8 cycles;
  * Carboplatin (AUC4) plus Gemcitabine 1000mg/m2 on day 1, 8 every 21 days for a maximum of 8 cycles;
  * Carboplatin (AUC5) plus Paclitaxel (175mg/m2) every 21days for a maximum of 8 cycles
  Arms: Chemotherapy

SUMMARY:
MITO 35b is designed as randomized, open label, phase III trial that aims to assess the efficacy of olaparib maintenance beyond progression compered to standard platinum-based chemotherapy after secondary cytoreductive surgery.

The target population of this study are ovarian cancer patients who experience a disease recurrence or progression to a first line maintenance therapy with PARPi; at progression patients must have received a secondary cytoreduction according to clinical practice.

ELIGIBILITY:
* Signed informed consent prior to any study specific procedures;
* Female, age ≥ 18 years at time of signing informed consent
* Patients with high-grade serous or endometroid ovarian, fallopian tube, or primary peritoneal cancer recurrent or progressive after first line PARPi maintenance are allowed;
* Patients must have received only one previous line of a platinum containing regimen not containing bevacizumab;
* Patient must have received a first-line maintenance therapy with a PARPi for at least 6 months, if the prior PARPi used was olaparib then patients must have received treatment without significant toxicity or the need for a permanent dose reduction.Patients who experience disease relapse after the end of the 24 months maintenance therapy are eligible;
* Patients must have undergone secondary cytoreductive surgery. The cytoreduction must result in complete resection (absence of macroscopic residual tumor) or at least resection of the progressive lesion(s) occurring during maintenance;
* Documented BRCA1/2 status. Both mutated and wild type patients are eligible. Patient with unknown status of BRCA genes agrees to undergo analysis of their germline and somatic BRCA status (testing must be completed prior to enrolment in the study);
* Patients must have a life expectancy ≥ 16 weeks;
* Patients must start the experimental treatments in the current study within 3 to 8 weeks from second surgery;
* ECOG performance status 0 to 1;
* Patient must provide archival tumor samples formalin fixed, paraffin embedded (FFPE) from both the primary and secondary surgeries for paired analysis. A quality control analysis of samples will be performed before patient's randomization;
* Patient must be able to take oral medications;
* Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

  * Haemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Total serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) and Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x ULN for the institution (or ≤ 5x ULN if liver metastases are present)
  * Patients must have creatinine clearance estimated of ≥51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test: Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F)a serum creatinine (mg/dL) x 72 (a where F=0.85 for females.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on Day 1 Cycle 1. Postmenopausal is defined as:

  * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50;
  * radiation-induced oophorectomy with last menses >1 year ago;
  * chemotherapy-induced menopause with >1-year interval since last menses;
  * surgical sterilisation (bilateral oophorectomy or hysterectomy).
* Women of childbearing potential and their partners, who are sexually active, must agree to the use of one highly effective forms of contraception and their partners must use a male condom, during the treatment and for at least 1 months after last dose of olaparib.For chemotherapy drugs, please refer to fertility section of corresponding Summary of Product Characteristics (SCP);
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures;

Exclusion Criteria:

* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, and/or active, uncontrolled infection. that may interfere with planned treatment, affect patient compliance or place the patient at high risk from treatment related complications [Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, New York Heart Association (NYHA) grade II or greater congestive heart failure, uncontrolled hypertension, severe peripheral vascular disease, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric illness ];
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication;
* Patients eligible for a platinum based chemotherapy doublet and bevacizumab;
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatments; prior palliative radiation must have been completed at least 7 days prior to the start of study drugs, and patients must have recovered from any acute adverse effects prior to the start of study treatment;
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of major surgery;
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT);
* Breast feeding women;
* Patients with symptomatic uncontrolled brain metastases. A TC/RMN scan of brain is required at baseline. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days;
* Other malignancy unless curatively treated with no evidence of disease for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS) and Stage 1, grade 1 endometrial carcinoma;
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable) except for transfusion done during surgery;
* Persistent toxicities >grade 2 according Common Terminology Criteria for Adverse (CTCAE) version 5.0 caused by previous cancer therapy, excluding alopecia;
* Resting ECG indicating uncontrolled, potentially irreversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation > 470 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome;
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks;
* Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents;
* Patients with myelodysplastic syndrome (MSD)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML;
* Immunocompromised patients, e.g., patients who are known to be serologically positive (HIV 1-2 antibody positivity) for human immunodeficiency virus (HIV);
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product;
* Patients that, at the Investigator's opinion, are not eligible according to ESMO (European society for Medical Oncology) guidelines for a re-treatment with a platinum containing therapy (i.e. patient has experienced a major adverse reaction to platinum salts during first line therapy);
* Patients with known active hepatitis (i.e. Hepatitis B or C)

  * Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Participation in another clinical study with an investigational product during the last 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2028-01-21 (Estimated); Study Completion 2028-01-21 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | until progression disease ( up to 5 years )
  PFS as defined by the Investigator using RECIST 1.1, as the time frame from randomization to progression or death for any cause,whichever comes first
Progession free survival 2 (PFS2) | until progression disease ( up to 5 years )
  PFS as defined by the Investigator using RECIST 1.1, as the time frame from randomization to second progression or death for any cause

SECONDARY OUTCOMES:
Overall survival | 5 years
  OS as defined by the Investigator as the time from randomization to death for any cause, whichever comes first.
Determination of changes in quality of life | At baseline, at Day 1 of each Cycle (during treatment) until 6 months, then at 9 and 12 months (up to 12 months).Each cycle is 28 days
  EORTC QLQ-C30, a quality questionnaire, composed by 30 items graded from 1 (not at all) to 4 (very much).
Determination of changes in patient-reported outcome (PRO) symptomatic toxicities | At baseline, at Day 1 of each Cycle (during treatment) until 6 months, then at 9 and 12 months (up to 12 months. Each cycle is 28 days
  PRO-CTCAE questionnaire, composed by 78 items graded from 1 (not at all) to 5 (very much).
Changes in patient-reported outcome (PRO) of cancer-related financial toxicity | t baseline, at day 1 of each Cycle (during treatment) until 6 months, then at 9 and 12 months (up to 12 months). Each cycle is 28 days
  The PROFFITquestionnaire consists of 16 items,graded from 1 (not at all) to 4 (very much).
Number of participants with treatment-related side effects | At baseline, day 1 of each cycle until progression disease (up to 5 years)].Each cycle is 28 days.
  Number of participants with treatment-related side effects
  Number of participants with treatment-related side effects graded according to Common Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Nazionale Tumori di Napoli, Naples, Italy

REFERENCES:
- [Derived] Schettino C, Musacchio L, Bartoletti M, Chiodini P, Arenare L, Baldassarre G, Califano D, Capoluongo E, Costi MP, D'Incalci M, Marchini S, Mezzanzanica D, Normanno N, Scala S, Greggi S, Perrone F, Pignata S. Olaparib beyond progression compared with platinum chemotherapy after secondary cytoreductive surgery in patients with recurrent ovarian cancer: phase III randomized, open-label MITO 35b study, a project of the MITO-MANGO groups. Int J Gynecol Cancer. 2022 Jun 6;32(6):799-803. doi: 10.1136/ijgc-2022-003435. PMID 35318277
- See also: Sponsor web-site for study conduction — https://usc.istitutotumori.na.it